CLINICAL TRIAL: NCT00319943
Title: Computer-Based Therapy for Mild Cognitive Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of California, San Francisco (Other); University of California, Davis (Other); Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OUT-108-2005
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2006-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive remediation; Cognitive impairment; computer; training
MeSH Terms: conditions — Cognitive Dysfunction

INTERVENTIONS:
Procedure: Computer-based training for Mild Cognitive Impairment (MCI)

SUMMARY:
The purpose of this study is to determine the neuropsychological and neurophysiological impacts of a computer-based training program designed to improve the cognitive performance of patients with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
The study is a randomized, double-blind, controlled trial of a computerized, cognitive intervention with three main goals: 1) to assess the magnitude of improvements in memory, language function, and cognitive function following computer training, 2) to investigate the neurophysiological mechanisms underlying such neuropsychological improvements, and 3) to demonstrate the feasibility of using this kind of computer-based therapy in older populations.

ELIGIBILITY:
Inclusion Criteria:

1)65 - 90 years of age 2)Meet definition for MCI including complaints of cognitive decline as indicated by patient report and/or informant report, and corroborated by clinician judgment and, the absence of dementia, defined as impairment of memory and at least one other domain of cognitive function.

3)Fluency in English 4)Willing to meet the time commitment of the study

-

Exclusion Criteria:

1. Clinically significant cerebrovascular disease
2. Individuals scheduled to begin acetylcholinesterase inhibitor (AChEI) therapy -

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48
Dates: Start 2004-09; Study Completion 2006-07

PRIMARY OUTCOMES:
The study investigates changes in a neuropsychological assessment battery pre-randomization
and upon the completion of training.

SECONDARY OUTCOMES:
Early evaluations will be conducted from brain imaging; specifically, date
obtained via positron emission tomography (PET), magnetoencephalography (MEG),
electroencephalography (EEG), and functional magnetic resonance imaging (fMRI)
studies.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Kramer, PsyD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Mejia AA, Nakamura T, Masatoshi I, Hatazawa J, Masaki M, Watanuki S. Estimation of absorbed doses in humans due to intravenous administration of fluorine-18-fluorodeoxyglucose in PET studies. J Nucl Med. 1991 Apr;32(4):699-706. PMID 2013810
- [Derived] Barnes DE, Yaffe K, Belfor N, Jagust WJ, DeCarli C, Reed BR, Kramer JH. Computer-based cognitive training for mild cognitive impairment: results from a pilot randomized, controlled trial. Alzheimer Dis Assoc Disord. 2009 Jul-Sep;23(3):205-10. doi: 10.1097/WAD.0b013e31819c6137. PMID 19812460